CLINICAL TRIAL: NCT00622713
Title: A 24 Week, Multicenter, Open, Evaluation of the Clinical Effectiveness of the Once-daily 10 cm2 Rivastigmine Patch Formulation in Patients With Probable Alzheimer's Disease (MMSE 10-26)
Brief Title: A 24 Week, Multicenter, Open, Evaluation of the Clinical Effectiveness of the Once-daily 10 cm^2 Rivastigmine Patch Formulation in Patients With Probable Alzheimer's Disease (EXTRA)
Acronym: EXTRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CENA713DFR08; N° EudraCT : 2007-003405-27
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Results first posted 2011-07-26 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-06

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; cholinesterase inhibitor; rivastigmine
MeSH Terms: conditions — Alzheimer Disease | interventions — Rivastigmine

INTERVENTIONS:
Drug: Rivastigmine transdermal patch — The study treatment was delivered as a patch sizes 5 and 10 cm^2 containing respectively 9 and 18 mg of rivastigmine. During the first 4 weeks of the study, patients applied a new rivastigmine 5 cm^2 patch once daily. At the end of the 4 weeks, if tolerability was satisfactory, the dosage was increased and patients applied rivastigmine 10 cm^2 patch once daily for an additional 4 weeks. Thereafter, and until the end of the study, patients remained at the maximum tolerated dose, either 5 or 10 cm^2.
  Other Names: Exelon, Prometax

SUMMARY:
This study is designed to confirm the efficacy, the tolerability, the patient compliance and the caregiver satisfaction with rivastigmine target patch size 10 cm^2 in patients with probable Alzheimer's Disease (Mini-Mental State Examination 10-26) in the community setting

ELIGIBILITY:
Inclusion Criteria:

* Males, and females of at least 50 years old with a primary caregiver
* Probable Alzheimer's disease
* Mini-Mental State Examination (MMSE) score of ≥ 10 and ≤ 26
* Patients initiating therapy for the first time with a Cholinesterase (ChE) inhibitor (patients prescribed both rivastigmine and memantine are allowed) or patients who failed to benefit from previous ChE inhibitor treatment
* Residing with someone in the community throughout the study or, if living alone, in contact with the responsible caregiver everyday

Exclusion Criteria:

* Patients not treated according to the product monograph for capsules
* Current diagnosis of an active skin lesion/disorder that would prevent accurate assessment of the adhesion and potential skin irritation of the patch (e.g., atopic dermatitis, wounded or scratched skin in the area of the patch application)
* History of allergy to topical products containing any of the constituents of the patches

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma S.A.S., Principal Investigator — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Rueil-Malmaison, France

RESULTS

PARTICIPANT FLOW:
Groups:
- Rivastigmine Transdermal Patch: During the first 4 weeks of the study, patients applied a new rivastigmine 5 cm^2 patch once daily. At the end of the 4 weeks, if tolerability was satisfactory, the dosage was increased and patients applied rivastigmine 10 cm^2 patch once daily for an additional 4 weeks. Thereafter, and until the end of the study, patients remained at the maximum tolerated dose, either 5 or 10 cm^2.
Period: Overall Study
Arm/Group | Rivastigmine Transdermal Patch
Started | 228
Exposed to Study Drug | 226
Intent to Treat (ITT) Population | 218
Completed | 169
Not Completed | 59
Not completed — Adverse Event | 35
Not completed — Administrative problems | 4
Not completed — Withdrawal by Subject | 11
Not completed — Lost to Follow-up | 5
Not completed — Death | 2
Not completed — Subject no longer required study drug | 1
Not completed — Did not meet eligibility criteria | 1

BASELINE CHARACTERISTICS:
Arm/Group | Rivastigmine Transdermal Patch
Number analyzed (Participants) | 218
Age Continuous [Mean (Standard Deviation); unit: years] — Baseline Measures are provided for the ITT population.
  years | 78.7 (6.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131
  Male | 87
Region of Enrollment [Number; unit: participants]
  France | 218

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Achieved and Maintained the Maximum Dose of 10 cm^2 Rivastigmine Patch for at Least 8 Weeks During 24 Weeks Study
Description: The primary endpoint was the percentage of patients who were able to tolerate (and stay on for at least 8 weeks) rivastigmine target patch size 10 cm^2.
Time Frame: 24 weeks
Population: The Intent-to-Treat (ITT) population was defined as all patients who were administered at least one dose of study medication and were assessed for efficacy at least 1 time.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivastigmine Transdermal Patch
Number analyzed (Participants) | 218
Percentage of participants | 70.6

2. Secondary Outcome: Clinical Global Impression of Change (CGI-C) by Physician
Description: The CGIC is an assessment tool used by a clinician to make a judgment of the severity or a change of a patient's condition. The clinician relies solely on information obtained from the patient at the Baseline visit as well as clinical information obtained throughout the study period. The CGIC is rated on the following seven-point scale:"very much improved", "much improved", "slightly improved", "unchanged", "slightly worsened", "much worsened" and "very much worsened".
Time Frame: Baseline and week 24
Population: The Intent-to-Treat (ITT) population was defined as all patients who were administered at least one dose of study medication and were assessed for efficacy at least 1 time. Last observation carried forward (LOCF) was used for missing values.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivastigmine Transdermal Patch
Number analyzed (Participants) | 208
Percentage of participants
  Very much improved | 4.3 (5.2)
  Much improved | 13.0
  Slightly improved | 23.1
  Unchanged | 32.2
  Slightly worsened | 19.2
  Much worsened | 5.8
  Very much worsened | 2.4

3. Secondary Outcome: Mean Change From Baseline to Week 24 in the 4-item Instrumental Activities of Daily Living (4-IADL) Score
Description: The 4-IADL assesses the ability of a patient to autonomously perform 4 activities of daily living: Use the telephone, take medications, use public transport, and manage their own budget. Each activity is assessed by a series of questions and rated on a scale of 1 to 4. Scores on the 4 activities are combined for a total score ranging from 1 to 16. A lower score indicates a more self-sufficient individual. A positive change from baseline score indicates worsening.
Time Frame: Baseline to week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rivastigmine Transdermal Patch
Number analyzed (Participants) | 218
scores on a scale
  Baseline (n= 198) | 3.2 (1.18)
  Week 24 (n= 181) | 3.2 (1.16)
  Change from Baseline to week 24 (n= 172) | 0.1 (0.74)

4. Secondary Outcome: Mean Change From Baseline to Week 24 in the Mini-Mental State Examination (MMSE) Score
Description: The MMSE is a brief, practical screening test for cognitive dysfunction. The test consists of five sections (orientation, registration, attention-calculation, recall, and language) and results in a total possible score from 0 to 30, with higher scores indicating better function. A positive change score indicates improvement from baseline.
Time Frame: Baseline to week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rivastigmine Transdermal Patch
Number analyzed (Participants) | 218
scores on a scale
  Baseline (n = 216) | 19.2 (4.11)
  Week 24 (n = 203) | 19.2 (5.19)
  Change from baseline to week 24 (n = 203) | 0.0 (3.18)

5. Secondary Outcome: Mean Change From Baseline to Week 24 in the Mini-Zarit Inventory Score
Description: The Mini-Zarit Inventory assesses the burden of a caregiver in caring for a patient. The inventory is composed of 5 questions which are rated according to the following answers: 0 = never, ½ = sometimes, 1 = often. The ratings on the 5 questions are added together resulting in a total score of 0 to 7 with a higher score indicating greater caregiver burden.
Time Frame: Baseline to week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Rivastigmine Transdermal Patch
Number analyzed (Participants) | 218
Scores on a scale
  Baseline (n= 211) | 2.8 (1.76)
  Week 24 (n= 199) | 2.9 (1.85)
  Change from baseline to week 24 (n= 197) | 0.1 (1.35)

ADVERSE EVENTS:
Description: Safety population.
Arm/Group | Rivastigmine Transdermal Patch
Serious Adverse Events (participants affected / at risk) | 21/218
Other Adverse Events (participants affected / at risk) | 13/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivastigmine Transdermal Patch (N=218)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1
BRADYCARDIA (Cardiac disorders) | 2
CARDIAC ARREST (Cardiac disorders) | 1
NAUSEA (Gastrointestinal disorders) | 1
SIGMOIDITIS (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 1
MALAISE (General disorders) | 1
OEDEMA PERIPHERAL (General disorders) | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 1
HEPATOMEGALY (Hepatobiliary disorders) | 1
HYPERSENSITIVITY (Immune system disorders) | 1
BRONCHITIS (Infections and infestations) | 1
LUNG INFECTION (Infections and infestations) | 1
VIRAL INFECTION (Infections and infestations) | 1
FALL (Injury, poisoning and procedural complications) | 5
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 1
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1
BIOPSY PROSTATE (Investigations) | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PROSTATIC ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
AUTONOMIC NERVOUS SYSTEM IMBALANCE (Nervous system disorders) | 1
DYSSTASIA (Nervous system disorders) | 1
EPILEPSY (Nervous system disorders) | 1
APATHY (Psychiatric disorders) | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 1
RASH (Skin and subcutaneous tissue disorders) | 1
SOCIAL STAY HOSPITALISATION (Social circumstances) | 1
HIP ARTHROPLASTY (Surgical and medical procedures) | 1
MALIGNANT TUMOUR EXCISION (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rivastigmine Transdermal Patch (N=218)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.